CLINICAL TRIAL: NCT06170554
Title: Study of Hydration Levels in Sports and Non-sports Schoolchildren
Brief Title: Study of Hydration Levels in Sports and Non-sports Schoolchildren (EHC)
Acronym: EHC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0201 - EHC
Record Dates: First submitted 2023-11-23; First posted 2023-12-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-12

CONDITIONS: Hydration
Keywords: Water; Beverage; Sports; Children; Middle school students; Adolescents; dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New knowledge regarding the negative impact of poor hydration on health highlights the need to provide recent epidemiological data on the water intake of the French population, especially among middle school students, a group that has been minimally studied until now. Given the crucial role of adequate hydration in sports performance, it is essential to assess fluid intake and hydration habits among middle school students, who often engage in intense physical activities. The primary outcome of this study is to evaluate whether the proportion of middle school students hydrating adequately according to current recommendations is higher among those engaging in moderate to intense sports compared to those who do little or no sports. The goal is to determine if daily fluid intake is significantly influenced by physical activity among this population. To achieve this, investigators have developed a questionnaire to gather information on the physical activity levels of middle school students, their daily hydration habits, and their liquid intake in relation to their sports activities, using appropriate visuals. This study involves distributing the questionnaire in two middle schools in Brittany between November 2023 and January 2024.

ELIGIBILITY:
Inclusion Criteria:

* Middle school students with little or no sports involvement and middle school students with a moderate to intense level of physical activity

Exclusion Criteria:

* Refusal of the middle school student to participate and parental opposition to their child's participation in this research

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The studied population includes middle school students from two classes of 6th, 5th, 4th, and 3rd grades at Sainte Anne College in Brest, as well as middle school students from two classes of 6th, 5th, 4th, and 3rd grades at Pays des Abers College in Lannilis.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of middle school students adhering to current hydration recommendations among both athletic and non-athletic middle school students | baseline
  Response to the questionnaire

SECONDARY OUTCOMES:
Proportion of middle school students adhering to current hydration recommendations | baseline
  Response to the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Agnes Giroux-Metges, MD PhD, Principal Investigator — Universitary Hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement